CLINICAL TRIAL: NCT06004102
Title: Impact of Text Message Reminders on Immunosuppressive Medication Adherence Among Kidney Transplant Recipients: A Randomized Controlled Study
Brief Title: Medication Adherence in Kidney Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University Hospital (Other)
Responsible Party: Principal Investigator, Kübra Erdal, Nurse, Akdeniz University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAEK-315
Record Dates: First submitted 2023-08-10; First posted 2023-08-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Medication Adherence
Keywords: kidney transplantation; reminder text messages; medication adherence; surgical nursing
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reminder text message (Experimental): At the baseline of the study, the Sociodemographic and Descriptive Characteristics Form and IMAS were administered to patients in the intervention groups as a pretest. Short text messages to remind the use of immunosuppressive medication and educational text messages were sent to patients in the intervention group four times a day, every day for three months. The intervention group also received educational text messages three days a week, in addition to such text message reminders.
  The text message contents prepared for the intervention group were sent automatically to patients at specified times via the purchased program. At the end of the study, intervention groups of participants completing the 9-month follow-up were administered the IMAS questionnaire as a posttest.
  Interventions: Other: reminder text message
- no intervention (No Intervention): At the baseline of the study, the Sociodemographic and Descriptive Characteristics Form and IMAS were administered to patients in the control groups as a pretest. The control group did not receive any such intervention. At the end of the study, control groups of participants completing the 9-month follow-up were administered the IMAS questionnaire as a posttest.

INTERVENTIONS:
Other: reminder text message — The study aimed to assess the impact of text message reminders on medication adherence among kidney transplant recipients.
  Arms: reminder text message

SUMMARY:
Aims and Objective: The study aimed to assess the impact of text message reminders on medication adherence among kidney transplant recipients.

Background: One of the most common problems encountered in transplant patients is incompatibility with immunosuppressive drugs, one of the most important reasons for graft rejection.

Design: A randomized controlled trial was conducted from January to October 2021 and conducted in accordance with the Consolidated Standards of Reporting Trials 2010 guidelines.

Methods: This randomized controlled trial included a total of 100 patients receiving a kidney transplant, 50 in the intervention group and 50 in the control group. Patients in the intervention group were sent text message reminders four times a day during the 6th to 9th months after transplantation. Control patients received no such intervention. Tacrolimus concentrations in the bloodstream were monitored for all participants through measurements taken at months 7,8, and 9. Data collection tools included Sociodemographic and Descriptive Characteristics Form and Immunosuppressive Medication Adherence Scale.

Research hypotheses H1- Sending text message reminders improves immunosuppressive medication adherence in kidney transplant recipients.

H2- Utilization of text messages as reminders has a significant influence on tacrolimus blood profiles in kidney transplant recipients.

H3- There is a correlation between the scores from the Immunosuppressive Medication Adherence Scale and mean tacrolimus plasma levels in kidney transplant recipients.

H4- There is a correlation between the sociodemographic and descriptive characteristics of kidney transplant recipients and their mean scores from the Immunosuppressive Medication Adherence Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Being a recipient of a kidney transplant for the first time
* Being a kidney transplant recipient at post-transplant month 6 with scheduled follow-up until month 9
* Ongoing immunosuppressive drug therapy
* Absence of any disability that hinders communication
* No diagnosis of psychological and mental problems
* Being an active cell phone user
* Ability to read and write
* Voluntary participation in the research.

Exclusion Criteria:

* Hospitalization for any reason during the research period
* History of combined or dual organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
The effect of sending reminder text messages on immunosuppressive medication adherence | baseline and 9 months
  The IMAS is a validated an 11-item self-report questionnaire developed in 2015 to measure medication adherence in patients that have received solid organ transplants and are prescribed immunosuppressive drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Konyaalti, Turkey (Türkiye)